CLINICAL TRIAL: NCT03445104
Title: Effect of Huperzine A on Cognitive Function and Perception of Effort During Exercise
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Chad Wessinger, BS, Graduate Assistant, St. Louis University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 28661
Record Dates: First submitted 2018-01-26; First posted 2018-02-26 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Cognitive Enhancement During Exercise
Keywords: Huperzine A; acetylcholinesterase inhibitor; AChEI; exercise; Physical performance; cognitive function; rating of perceived exertion; RPE
MeSH Terms: conditions — Motor Activity | interventions — huperzine A

STUDY DESIGN:
Intervention Model Description: The participants will be randomized to receive huperzine A or placebo during the first session. They will then receive the other treatment during the second session.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization allocation will be performed by personnel not involved in data collection to maintain participant and investigator blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huperzine A (Experimental): Huperzine A will be provided in the form of a single capsule for oral ingestion.
  Interventions: Other: Huperzine A
- Rice Flour (Placebo Comparator): Placebo will be provided in the form of a single capsule for oral ingestion.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Huperzine A — During one of the two experimental sessions, participants will be given huperzine A.
  Arms: Huperzine A
Other: Placebo — During one of the two experimental sessions, participants will be given a placebo.
  Arms: Rice Flour

SUMMARY:
This study evaluates the effects of acute huperzine A ingestion prior to exercise on cognitive function and perceived effort in exercise-trained individuals. Huperzine A has shown the ability to improve cognitive function in dementia patients, and is currently marketed as a cognitive enhancing supplement. Study participants will receive either huperzine A or placebo during the first experimental session, and will receive the other substance during the second session.

DETAILED DESCRIPTION:
Huperzine A improves cognitive function by inhibiting the enzyme acetylcholinesterase. This enzyme is responsible for the degradation of the neurotransmitter acetylcholine. inhibition of acetylcholinesterase may allow for greater availability of acetylcholine, which may allow for better nerve conduction and therefore enhanced cognitive function and possibly muscular contraction.

Huperzine A (200 mcg, Swanson®, Fargo, North Dakota) and placebo capsules will be administered in a single oral dose. The dose of Huperzine A to be used is comparable to previous research (Xu et al, 2011). Placebo capsules will consist of rice flour. The participants will ingest the capsules with 250 mL of water 30-45 minutes before exercise is initiated.

A paired-sample t-test with alpha set to p ≤ 0.05 for statistical significance will be used to analyze the data. Outcomes measured during the first and second experimental sessions will be compared to each other. The participants will be compared to themselves during previous sessions, so a paired sample t-test will be used to calculate the difference between the sessions. Data will be presented as means ± SE. Data analyses will be performed with Microsoft Excel; and other analyses may be performed as needed to gain further insights about the data.

A statistical power analysis was performed (G*Power software, version 3.1.5, University of Kiel, University of Dusseldorf, and University of Mannheim, 157 Germany) based on the following inputs: two-tailed paired t-test, alpha=0.05, desired power=0.80, sample size=15 subjects. The results indicated that a standardized effect size of 0.78 (i.e. large effect) will be detectable. As many as 20 subjects will be recruited and enrolled to ensure that complete data on 15 subjects are available in the event of screen fails and dropouts.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of all ethnic and racial groups that participate in endurance exercise of moderate to vigorous intensity at least three days per week, for at least 20 minutes per session, for at least six months prior to this study

Exclusion Criteria:

* Anyone not within the age range listed in section 8a will be excluded. Individuals who require medical clearance to participate in vigorous exercise based on ACSM's risk assessment algorithm will be excluded from the study. The participant screening form will be used to identify signs and symptoms or medical conditions that require medical clearance to participate in vigorous exercise.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Digit span | This test will be implemented during a 2 minute window during the last 10 minutes of endurance exercise.
  Digit span will be used as a measure of working memory. During a period of two minutes, the participants will be presented with a series of digits at a rate of one digit per second, and will be required to to repeat them verbatim. If they succeed, they will be presented with a longer series by one digit. The longest series that they are able to correctly repeat will be the number of their score (i.e. if they are able to repeat a series of 7 digits, their score will be 7).
Verbal Fluency | This test will be implemented during a 1 minute window during the last 10 minutes of endurance exercise.
  Verbal fluency will be used as a measure of executive function. Participants will be instructed to generate words beginning with F, A, S, B, H, or R. Each participant will be randomly assigned a different letter at each session.
Category Fluency | This test will be implemented during a 1 minute window during the last 10 minutes of endurance exercise.
  Category fluency will be used as a measure of executive function. Participants will be instructed to produce as many words as they can for a particular category within one minute. Each participant will be randomly assigned a different category at each session.
Stroop Effect Test | This test will be implemented during a 2 minute window during the last 10 minutes of endurance exercise.
  The Stroop effect test will be used as a measure of information processing. Participants will be exposed to color names printed in an ink color that does not match the color name. They will be instructed to name the color of the ink and to ignore the color name.

CONTACTS AND LOCATIONS:
Locations (1):
- Allied Health Professional Building, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided